CLINICAL TRIAL: NCT00450320
Title: A Pilot Study of Rapamycin in Patients With HIV-Related Kaposi's Sarcoma
Brief Title: Sirolimus in Treating Patients With HIV-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-051; U01CA070019 (NIH); CDR0000536481 (Other: NCI); WYETH-0468X-4420 (Other: Wyeth)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Sarcoma
Keywords: AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma
MeSH Terms: conditions — Sarcoma; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rapamycin (Active Comparator): The target rapamycin trough level will be 5-10 ng/mL. The initial dose will be dependent upon the type of HAART regimen.
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: sirolimus — The target rapamycin trough level will be 5-10 ng/mL. The initial dose will be dependent upon the type of HAART regimen. Subjects will continue on study protocol for six cycles as long as their KS is stable or continuing to respond to study medication. Treatment will be extended for up to six additional cycles if the subject has met criteria for a response. Subjects with no more than stable disease will have treatment discontinued after six cycles. Protocol treatment will be discontinued if the subject develops tumor progression, unacceptable toxicity or develops one of the protocol-defined reasons for treatment discontinuation at any time during the study.
  Other Names: rapamycin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as sirolimus, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sirolimus also may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This pilot study is studying sirolimus in treating patients with HIV-related Kaposi's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and toxicity of sirolimus in patients with HIV-related Kaposi's sarcoma (KS) receiving protease inhibitor (PI)-based or nonnucleoside reverse transcriptase inhibitor (NNRTI)-based highly active antiretroviral treatment (HAART) regimens.
* Estimate the dose(s) of this drug required to achieve target trough sirolimus plasma concentrations of 5-10 ng/mL in patients receiving PI-based or NNRTI-based HAART regimens.

Secondary

* Evaluate the clinical response of KS in patients treated with this sirolimus.
* Determine the effects of this drug on mTOR-dependent signaling in peripheral blood mononuclear cells (PBMC) and KS tumor biopsies.
* Determine the serum cytokine profiles pre- and post-treatment with this drug.
* Determine the effects of this drug on HIV and KS-associated herpesvirus (KSHV) viral loads.
* Determine the effects of this drug on T-lymphocyte subsets.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 3 treatment groups.

* Group 1 (patients receiving PI-based HAART regimen with ritonavir): Patients receive oral sirolimus 0.0015 mg/kg/day once daily on days 1-28 for 6 courses as long as KS is stable or the disease is continuing to respond to treatment. Patients may receive 6 additional courses provided they meet criteria for response in the absence of disease progression or unacceptable toxicity. Patients with no more than stable disease after 6 courses are discontinued from treatment.
* Group 2 (patients receiving PI-based HAART regimen without ritonavir): Patients receive oral sirolimus 0.003 mg/kg/day as in group 1.
* Group 3 (patients receiving NNRTI-based HAART regimen): Patients receive oral sirolimus 0.05 mg/kg/day as in group 1.

Blood samples are collected periodically and analyzed for sirolimus levels via LCMSMS.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven Kaposi's sarcoma (KS) involving 1 or more of the following tissues:

  * Skin
  * Lymph nodes
  * Oral cavity
  * Gastrointestinal tract and/or lungs, if the disease meets the following criteria:

    * Asymptomatic or minimally symptomatic
    * Require systemic cytotoxic therapy
* At least five measurable, previously non-irradiated, cutaneous lesions (indicator lesions)

  * Three non-indicator cutaneous lesions ≥ 4 x 4 mm accessible for 3-mm punch biopsy
* Serologic documentation of HIV infection (i.e., positive enzyme-linked immunosorbent assay, positive western blot, or other federally approved licensed HIV test, or a detectable blood level of HIV RNA)

  * CD4 count > 50 cells/µL
  * Serum HIV RNA level < 400 copies/mL
* KS that is either stable or progressing in the 4 weeks prior to study entry after being on stable antiretroviral therapy for ≥ 12 weeks with a PI-based or NNRTI-based regimen of ≥ 3 drugs, with no intention to change the regimen within 8 weeks of starting study drug

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy ≥ 3 months
* Hemoglobin ≥ 8.0 g/dL
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 75,000/mm³
* Glomerular filtration rate > 40 mL/min
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) (≤ 3.5 mg/dL if due to indinavir therapy and direct bilirubin normal; no limit if due to atazanavir therapy and direct bilirubin is normal)
* AST and ALT ≤ 2.5 times ULN
* Fasting triglyceride ≤ 400 mg/dL (4.5 mmol/L)
* Total cholesterol ≤ 300 mg/dL (7.8 mmol/L)
* Spot urine protein:creatinine ratio ≤ 0.5 and/or proteinuria ≤ 500 mg
* No other prior or concurrent malignancy except for treated basal cell skin cancer or carcinoma in situ of the cervix
* No evidence of infiltrate, cavitation, or consolidation (i.e., due to infection or other serious medical illness) on chest x-ray within the past 3 months
* No known hypersensitivity to sirolimus or its derivatives or macrolide antibiotics
* No New York Heart Association class III-IV cardiac disease (e.g., myocardial infarction within the past 6 months)
* No other concurrent severe and/or life-threatening medical disease
* No acute or known chronic liver disease (e.g., chronic active hepatitis or cirrhosis)

  * Hepatitis C with documentation of no or minimal fibrosis on liver biopsy allowed
* No concurrent active opportunistic infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier-method contraception during and for 3 months after completion of study therapy

PRIOR CONCURRENT THERAPY:

* No prior sirolimus
* No acute treatment for infection or other serious medical illness within the past 14 days
* No anticancer therapy for KS, including chemotherapy, radiotherapy, or biological therapy within the past 4 weeks (6 weeks for nitrosoureas or mitomycin C)
* No local therapy for any KS indicator lesion within the past 60 days, unless the lesion has progressed since treatment
* No investigational therapies within the past 4 weeks
* No major surgery within the past 2 weeks
* No prior or concurrent treatment with agents or medications, other than antiretroviral drugs used to treat HIV infection, that would interfere with the metabolism or excretion of sirolimus, including, but not limited to, the following:

  * Antifungals (e.g., voriconazole, itraconazole, or ketoconazole)
  * Antibiotics (e.g., erythromycin, telithromycin, clarithromycin, rifampin, or rifabutin)
  * Cidofovir
  * Cisapride
  * Diltiazem
  * Cyclosporine
  * Grapefruit juice
  * Hypericum perforatum (St. John's wort)
* No other concurrent anticancer therapies, including chemotherapy, biological therapy, or radiotherapy
* No concurrent systemic corticosteroid treatment, other than replacement doses
* No other concurrent investigational therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity | All study visits
Dose of sirolimus required to achieve target trough sirolimus plasma concentration | Days 8, 15, 21, 29, 43, 57, 85, 113, and every 28 days thereafter

SECONDARY OUTCOMES:
Clinical response | Days 1, 29, 57, 85, every 28 days thereafter, at treatment discontinuation, and at study discontinuation.
Effect of sirolimus on mTOR-dependent signaling in peripheral blood mononuclear cells (PBMC) and Kaposi's sarcoma (KS) tumor biopsies | baseline, days 1, 15, 29, 57, 113, every 28 days thereafter, study discontinuation
Serum cytokine profile | baseline, days 1, 15, 29, 57, 113, every 28 days thereafter, study discontinuation
Effect of sirolimus on HIV and KS-associated herpesvirus viral loads | Days 1, 15, 29, 57, 113, every 28 days thereafter, study discontinuation
Effect of sirolimus on T-lymphocyte subsets | Baseline, Days 29, 113, and at treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Susan E. Krown, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Dirk Dittmer, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York